CLINICAL TRIAL: NCT06974058
Title: Evaluation of a Quercetin/Curcumin-Based Supplement for Mild to Moderate Long COVID-19 Symptoms: A Pragmatic, Interventional Clinical Study.
Brief Title: Study to Investigate the Health Benefits of a Quercetin/Curcumin-Based Supplement for Mild to Moderate Long COVID-19 Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental medicine, Liaquat University of Medical & Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUMHS/REC/-735/13.05.2025
Record Dates: First submitted 2025-05-12; First posted 2025-05-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Quercetin

STUDY DESIGN:
Intervention Model Description: This is a pragmatic, open-label clinical study evaluating the benefits of a combined quercetin/curcumin supplement (Nasafytol®) in adults experiencing mild to moderate Long COVID-19 symptoms.
Masking Description: None (Open Label) (Participants and researchers will be aware of the treatment)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nasafytol® Group (Quercetin/Curcumin Supplement Group) (Experimental): Participants in this group will receive a combined supplement of Nasafytol®, containing quercetin (65 mg) and curcumin (42 mg). Participants will be instructed to take two capsules (single administration) twice a day for 8 weeks.
  Interventions: Dietary Supplement: Nasafytol® (Quercetin/Curcumin Supplement)

INTERVENTIONS:
Dietary Supplement: Nasafytol® (Quercetin/Curcumin Supplement) — Participants in this group will receive Nasafytol®, a combined dietary supplement containing quercetin (65 mg) and curcumin (42 mg). Participants will take two capsules (single administration) twice a day for a duration of 8 weeks. The supplement is intended to alleviate mild to moderate symptoms of Long COVID-19, including but not limited to fatigue, cognitive function, generalized body pain, low mood, sleep disturbance, and overall quality of life.

SUMMARY:
This pragmatic clinical study aims to evaluate the efficacy and tolerance of a combined quercetin/curcumin supplement in adults experiencing mild to moderate symptoms of Long COVID-19. Participants will receive the combined quercetin/curcumin supplement for 2 months. The primary outcome is the improvement in overall symptom burden, while secondary outcomes include changes in quality of life, the need for NSAIDs, and inflammatory markers. The study seeks to provide real-world evidence of the potential benefits of this combined supplement in managing Long COVID-19 symptoms.

DETAILED DESCRIPTION:
Long COVID-19, characterized by persistent symptoms lasting weeks or months after the acute phase of SARS-CoV-2 infection, presents a significant challenge for healthcare systems and affected individuals. Common symptoms include fatigue, brain fog, muscle pain, joint pain, sleep disturbances, and generalized weakness. Despite extensive research, there are limited effective therapeutic options for managing Long COVID-19 symptoms.

Quercetin and curcumin, two natural compounds with well-documented anti-inflammatory, antioxidant, and immunomodulatory properties, have gained attention for their potential benefits in various inflammatory and infectious conditions. Quercetin, a flavonoid found in various fruits and vegetables, has been shown to inhibit pro-inflammatory cytokines, reduce oxidative stress, and modulate immune responses. Curcumin, a polyphenol derived from turmeric (Curcuma longa), is known for its strong anti-inflammatory and antioxidant properties and has demonstrated immune-modulating effects in clinical studies.

Nasafytol® is a standardized combination supplement containing bioactive quercetin (65 mg) and curcumin (42 mg) from Curcuma longa, specifically formulated to enhance bioavailability and provide synergistic benefits. Both quercetin and curcumin in Nasafytol® are optimized for absorption and efficacy, making it a promising intervention for managing inflammatory and immune-related conditions.

The combination of quercetin and curcumin in Nasafytol® is hypothesized to provide synergistic benefits in managing Long COVID-19 symptoms. This pragmatic clinical study aims to evaluate the efficacy of Nasafytol® in reducing symptom burden and improving quality of life in adults experiencing mild to moderate Long COVID-19 symptoms. Participants will receive the combined supplement for two months, with primary outcomes focused on symptom improvement and secondary outcomes assessing changes in quality of life, the need for NSAIDs, and inflammatory markers.

The study is designed as a real-world pragmatic trial to provide evidence of the potential health benefits of Nasafytol® for Long COVID-19, addressing a critical gap in current management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years.
* History of confirmed COVID-19 infection at least 6 months prior to the enrollment.
* Persistent mild to moderate COVID-19 symptoms for at least 3 months post-acute infection.
* Diagnosis of Long COVID-19 based on WHO criteria.
* Symptom burden score of ≥25 at baseline (V0) on the COVID-19 Yorkshire Rehabilitation Scale (C19-YRS).
* At least one symptom scoring between 1-7 on the C19-YRS.
* Stable medical condition: No recent hospitalization (past 3 months) due to acute illness.
* Willing and able to adhere to the study protocol, including follow-up visits, symptom reporting, and compliance with supplementation

Exclusion Criteria:

* Hypersensitivity or allergy to quercetin, curcumin, or any component of the supplement (Nasafytol®).
* Severe, uncontrolled chronic illness (e.g., severe heart failure, chronic kidney disease requiring dialysis, severe liver disease).
* Regular use of quercetin or curcumin supplements within the last 3 months.
* Use of anticoagulants (e.g., warfarin, heparin, DOACs) due to potential anticoagulant effects of quercetin/curcumin.
* Acute illness at the time of screening.
* Pregnancy or breastfeeding.
* Use of immunosuppressive medications or corticosteroids within the past month.
* Significant psychiatric disorder that may interfere with study compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2025-07-22 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-12-14 (Actual)

PRIMARY OUTCOMES:
Change in Overall Symptom Burden | 8 weeks
  Assessment of overall symptom burden using the COVID-19 Yorkshire Rehabilitation Scale (C19-YRS). Improvement will be defined as either a ≥2-point reduction in any single symptom domain or a ≥10% reduction in the total C19-YRS symptom burden score from baseline.

SECONDARY OUTCOMES:
Change in Functional Status and Quality of Life (SF-36 Scores) | 8 weeks
  Assessment of quality of life using the SF-36 Health Survey, which evaluates eight domains, including physical functioning, bodily pain, general health, vitality, social functioning, and emotional well-being. It provides two summary scores: physical and mental health components.
Change in the Need for Prescribed Medications or NSAIDs (Non-Steroidal Anti-Inflammatory Drugs) | 8 weeks
  Monitoring the frequency and dosage of prescribed medications or NSAIDs (Non-Steroidal Anti-Inflammatory Drugs) used for symptom relief. This will be recorded using a participant-maintained medication log.
Change in Pain Severity and Pain Interference (Brief Pain Inventory - Short Form) | 8 weeks
  The Brief Pain Inventory - Short Form (BPI-SF) is a validated, self-reported questionnaire that assesses the severity of pain and the impact of pain on daily functioning. The instrument includes items measuring pain intensity (worst, least, average, and current pain) and pain interference with general activity, mood, walking ability, normal work, relations with others, sleep, and enjoyment of life. Scores range from 0 to 10, with higher scores indicating greater pain severity or interference.
Change in Fatigue Severity (Fatigue Severity Scale) | 8 weeks
  The Fatigue Severity Scale (FSS) is a 9-item, self-administered questionnaire designed to assess the severity of fatigue and its impact on daily activities and functioning. Each item is rated on a 7-point Likert scale, with higher scores indicating greater fatigue severity.
Change in Anxiety and Depression Symptoms (Hospital Anxiety and Depression Scale) | 8 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a validated, 14-item self-report instrument used to assess symptoms of anxiety and depression. It consists of two subscales (anxiety and depression), each with 7 items. Subscale scores range from 0 to 21, with higher scores indicating greater symptom severity.
Change in Sleep Quality (Pittsburgh Sleep Quality Index) | 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a validated self-reported questionnaire that assesses sleep quality and sleep disturbances over a 1-month interval. It consists of 19 items generating seven component scores and a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality.
Change in Cognitive Function (PROMIS Cognitive Function - Short Form 8a) | 8 weeks
  The PROMIS® Cognitive Function - Short Form 8a is a validated, patient-reported outcome measure assessing perceived cognitive abilities, including memory, attention, and mental clarity. The instrument consists of 8 items and is scored using standardized T-scores, with higher scores indicating better cognitive function.

CONTACTS AND LOCATIONS:
Locations (1):
- Liaquat University of Medical & Health Sciences (LUMHS), Jamshoro, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vollbracht C, Kraft K. Oxidative Stress and Hyper-Inflammation as Major Drivers of Severe COVID-19 and Long COVID: Implications for the Benefit of High-Dose Intravenous Vitamin C. Front Pharmacol. 2022 Apr 29;13:899198. doi: 10.3389/fphar.2022.899198. eCollection 2022. PMID 35571085
- [Background] Vlaming-van Eijk LE, Bulthuis MLC, van der Gun BTF, Wold KI, Veloo ACM, Vincenti Gonzalez MF, de Borst MH, den Dunnen WFA, Hillebrands JL, van Goor H, Tami A, Bourgonje AR. Systemic oxidative stress associates with the development of post-COVID-19 syndrome in non-hospitalized individuals. Redox Biol. 2024 Oct;76:103310. doi: 10.1016/j.redox.2024.103310. Epub 2024 Aug 19. PMID 39163767
- [Background] Al-Hakeim HK, Al-Rubaye HT, Al-Hadrawi DS, Almulla AF, Maes M. Long-COVID post-viral chronic fatigue and affective symptoms are associated with oxidative damage, lowered antioxidant defenses and inflammation: a proof of concept and mechanism study. Mol Psychiatry. 2023 Feb;28(2):564-578. doi: 10.1038/s41380-022-01836-9. Epub 2022 Oct 24. PMID 36280755
- [Background] Gerain J, Uebelhoer M, Costes B, Herman J, Pietri S, Donneau AF, Monseur J, Henrotin Y. NASAFYTOL(R) supplementation in adults hospitalized with COVID-19 infection: results from an exploratory open-label randomized controlled trial. Front Nutr. 2023 Jun 22;10:1137407. doi: 10.3389/fnut.2023.1137407. eCollection 2023. PMID 37426178
- [Background] Khan A, Iqtadar S, Mumtaz SU, Heinrich M, Pascual-Figal DA, Livingstone S, Abaidullah S. Oral Co-Supplementation of Curcumin, Quercetin, and Vitamin D3 as an Adjuvant Therapy for Mild to Moderate Symptoms of COVID-19-Results From a Pilot Open-Label, Randomized Controlled Trial. Front Pharmacol. 2022 Jun 7;13:898062. doi: 10.3389/fphar.2022.898062. eCollection 2022. PMID 35747751
- [Background] Ujjan ID, Khan S, Nigar R, Ahmed H, Ahmad S, Khan A. The possible therapeutic role of curcumin and quercetin in the early-stage of COVID-19-Results from a pragmatic randomized clinical trial. Front Nutr. 2023 Jan 18;9:1023997. doi: 10.3389/fnut.2022.1023997. eCollection 2022. PMID 36742008